CLINICAL TRIAL: NCT04137783
Title: ABCA3 Gene Mutations in Late Preterm and Term Infants With Fatal Unexplained Respiratory Distress Syndrome
Brief Title: ABCA3 Gene and RDS in Late Preterm and Term Infants
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Wang Jianhui, Attending Doctor, Children's Hospital of Chongqing Medical University
Other Study IDs: 00020191017
Record Dates: First submitted 2019-10-20; First posted 2019-10-24 (Actual); Results first posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: respiratory distress syndrome; ABCA3 gene; exome sequencing
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- homozygous or compound heterozygous ABCA3 mutations: patients meet the criteria for fatal respiratory distress sydrome and undergone exome sequencing, which indicated homozgyous or compound heterozygous ABCA3 mutations.
  Interventions: Other: no intervention
- single ABCA3 mutation: patients meet the criteria for fatal respiratory distress sydrome and undergone exome sequencing, which indicated single mutations.
  Interventions: Other: no intervention
- no ABCA3 mutations: patients meet the criteria for fatal respiratory distress sydrome and undergone exome sequencing, which exclude all gene mutations involving in the respiratory disease.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — there is no intervention in this study, only observation.

SUMMARY:
Respiratory distress syndrome (RDS) is the most common respiratory cause of mortality and morbidity in very preterm infants, but it also could be seen in late preterm and term infants. Some genetic mechanisms were involved in the pathogenesis of RDS in late preterm and term infants.

ATP-binding cassette transporter A3 (ABCA3) is essential for the production of pulmonary surfactant, whose mutation is the most common monogenetic cause of RDS in newborns. It also takes a vital role on unexplained RDS (URDS) in late preterm and term infants. Some previous studies showed that URDS with homozygous or compound heterozygous ABCA3 mutations had high mortality, while different mutation types could lead to different outcomes. However, most of the study focused on URDS with ABCA3 gene mutations, and there is no evidence that URDS without confirmed gene mutations have relatively better or worse outcomes. Furthermore, all the population in previous study are non-Asian races, which indicated that all the study conclusion is not applicable in Asia.

Based on the next-generation sequencing technology, exome sequencing has been widely used in the clinic. In our neonatal intensive care unit (NICU), a clinic exome sequencing was usually performed in infants with fatal URDS. The present study was designed to compare the URDS with ABCA3 gene mutations with those without confirmed gene mutations and to establish the relationship between various ABCA3 gene mutations and variant RDS severity and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* infants ≥34 weeks' gestation
* meet the fatal respiratory distress syndrome as following: (1) manifestations and chest radiograph are compatible with RDS; (2) at least 7days on invasive ventilation with FiO2 ≥60%, or persistent hypoxemic respiratory failure on FiO2 100% regardless of duration of invasive ventilation
* undergone exome sequencing

Exclusion Criteria:

* culture-positive sepsis
* cardiopulmonary malformations
* pulmonary hypoplasia
* known surfactant mutations such as SFTPB, SFTPC, CHPT1, LPCAT1 and PCYT1B were excluded.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All the infants ≥34 weeks'gestation was admitted in neonatal intensive care unit of Children's Hospital of Chongqing Medical University from January 2013 to December 2018
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wang Jianhui, Doctor, Principal Investigator — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Homozygous or Compound Heterozygous ABCA3 Mutations | Single ABCA3 Mutation | no ABCA3 Mutations
Started | 7 | 10 | 22
Completed | 7 | 10 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Homozygous or Compound Heterozygous ABCA3 Mutations | Single ABCA3 Mutation | no ABCA3 Mutations | Total
Number analyzed (Participants) | 7 | 10 | 22 | 39
Age, Customized [Mean (Standard Deviation); unit: weeks]
  Gestational age | 36.85 (2.12) | 36.80 (1.81) | 37.27 (2.27) | 37.08 (2.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 10 | 18
  Male | 4 | 5 | 12 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 10 | 22 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Birthweight(grams) [Mean (Standard Deviation); unit: grams] | 2996.57 (351.92) | 2934.10 (517.68) | 3043.59 (358.03) | 3007.08 (395.04)
Cesarean section (n, %) [Count of Participants; unit: Participants] | 5 | 5 | 14 | 24
Resuscitation (n, %) [Count of Participants; unit: Participants] | 4 | 4 | 6 | 14
Fetal distress (n, %) [Count of Participants; unit: Participants] | 2 | 3 | 4 | 9
Meconium stained amniotic fluid (n, %) [Count of Participants; unit: Participants] | 2 | 2 | 3 | 7
Maternal history [Count of Participants; unit: Participants]
  premature rupture of membrane | 2 | 3 | 5 | 10
  gestational diabetes mellitus | 2 | 2 | 7 | 11
  Preeclampsia | 1 | 1 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: the ratio of dead patients against the corresponding group population
Time Frame: through study completion, an average of 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Homozygous or Compound Heterozygous ABCA3 Mutations | Single ABCA3 Mutation | no ABCA3 Mutations
Number analyzed (Participants) | 7 | 10 | 12
Participants | 5 | 3 | 5

2. Secondary Outcome: the Onset of Respiratory Distress Syndrome
Description: the age when the patients presented with respiratory distress sydnrome
Time Frame: up to 1 week
Measure: Mean (Full Range); unit: hours
Arm/Group | Homozygous or Compound Heterozygous ABCA3 Mutations | Single ABCA3 Mutation | no ABCA3 Mutations
Number analyzed (Participants) | 7 | 10 | 12
hours | 1.83 [0.1 to 5] | 4.6 [1 to 10] | 5.24 [0.1 to 13]

3. Secondary Outcome: the Age of Developing Severe RDS Marked With Oxygenation Index of 16
Description: the age when the patients develop severe RDS,which is marked with an oxygenation index of 16
Time Frame: through study of completion, an average of 1 month
Measure: Mean (Full Range); unit: days
Arm/Group | Homozygous or Compound Heterozygous ABCA3 Mutations | Single ABCA3 Mutation | no ABCA3 Mutations
Number analyzed (Participants) | 7 | 10 | 12
days | 1.06 [0.1 to 2] | 5.3 [2 to 15] | 4.5 [1 to 11]

4. Secondary Outcome: Radiological Score
Description: The chest x-ray was rated in three sections on both sides of the lung: apex to the carina, carina to the lower pulmonary vein, and lower pulmonary vein to diaphragm. The incidence of radiological features, including ground-glass opacity, reticular pattern, air bronchogram, atelectasis, and air leak, was evaluated for each lung section, respectively. Each finding was scored as 0=none, 1=discrete，2=diffuse, and 3= strong at each section. An overall cumulative score was calculated by adding the individual section scores together, making a minimum of 0, and a maximum of 18 for each patient. Higher scores mean the higher severity of the radiological apperance, and commonly predict worse respiratory outcomes.
Time Frame: through study of completion, an average of 1 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Homozygous or Compound Heterozygous ABCA3 Mutations | Single ABCA3 Mutation | no ABCA3 Mutations
Number analyzed (Participants) | 7 | 10 | 12
score on a scale
  ground glass opacity | 15.29 (1.38) | 12.90 (2.03) | 10.77 (1.95)
  reticular pattern | 15.14 (1.22) | 14.90 (0.88) | 13.23 (2.11)
  air bronchogram | 11.86 (2.34) | 11.00 (1.25) | 7.86 (3.09)
  atelectasis | 5.57 (2.82) | 3.20 (2.35) | 2.64 (0.91)
  air leakage | 1.43 (1.99) | 1.20 (1.40) | 0.91 (1.07)
  cysts | 1.86 (2.04) | 1.00 (1.25) | 0.50 (0.86)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 month
Arm/Group | Homozygous or Compound Heterozygous ABCA3 Mutations | Single ABCA3 Mutation | no ABCA3 Mutations
All-Cause Mortality (participants affected / at risk) | 5/7 | 3/10 | 11/22
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10 | 0/22
Other Adverse Events (participants affected / at risk) | 0/7 | 0/10 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT04137783/Prot_SAP_000.pdf